CLINICAL TRIAL: NCT03280017
Title: Low Dose Intraoperative Intravenous Ketamine in Combination With Multilevel Paravertebral Block for Post Video-assisted Thoracic Surgery Pain: a Randomized Study
Brief Title: Ketamine With Multilevel Paravertebral Block for Post Video-assisted Thoracic Surgery Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Sirilak Suksompong, Associate Professor, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 297/2560(EC1)
Record Dates: First submitted 2017-09-10; First posted 2017-09-12 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Pain, Acute; Pain, Chronic; Pain, Neuropathic
Keywords: anesthesia; thoracic surgery; thoracic paravertebral block; ketamine
MeSH Terms: conditions — Acute Pain; Chronic Pain; Neuralgia | interventions — Ketamine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketamine (Experimental): Participant allocated to this arm will receive intravenous ketamine infusion starting after the induction of anesthesia until the end of the surgery at the beginning of skin closure Participant will receive an ultrasound-guide thoracic paravertebral block using 0.5% plain bupivacaine prior to the induction of anesthesia
  Interventions: Drug: Ketamine
- Normal saline (Placebo Comparator): Participant allocated to this arm will receive intravenous normal saline solution infusion starting after the induction of anesthesia until the end of the surgery at the beginning of skin closure Participant will receive an ultrasound-guide thoracic paravertebral block using 0.5% plain bupivacaine prior to the induction of anesthesia
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Ketamine — intravenous ketamine 0.2 mg/kg/hr (concentration 1 mg/ml)
  Arms: Ketamine
Drug: Normal saline — normal saline infusion
  Arms: Normal saline

SUMMARY:
Postoperative pain after thoracic surgery is associated with adverse outcomes. The current strategy to prevent postoperative pain is the use of regional anesthesia and analgesic agents. In video-assisted thoracic surgery (VATS), thoracic paravertebral block has become the standard analgesic regimen which results in decreased postoperative pain and opioid consumption.

The investigator would like to study the analgesic efficacy of low dose intravenous ketamine infusion during surgery in combination with thoracic paravertebral block on postoperative pain after VATS in a randomized study.

DETAILED DESCRIPTION:
Inadequate pain control after thoracic surgery is associated with adverse events such as postoperative pulmonary complications (PPC), and chronic post surgical pain.

Although the less invasive video-assisted thoracic surgery (VATS) has been used extensively as it produces optimal surgical outcomes and possible less postoperative pain, there are reports of inadequate pain control.

Thoracic paravertebral block (TPVB) has been introduced as an effective method in postoperative pain management after VATS. It is associated with improved pain control and the reduction of opioid analgesic consumption in several studies.

The use of intravenous low dose ketamine infusion during and after surgery has been shown to produce superior postoperative pain control in upper abdominal surgery and thoracotomy.

The aim of the present study is to study the efficacy of intravenous low dose ketamine infusion during surgery on acute and chronic pain after VATS.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologist physical status 1-3
* Scheduled for elective video-assisted thoracic surgery
* Able to operate a patient-controlled analgesia device (PCA)

Exclusion Criteria:

* History of morphine allergy
* History of bupivacaine allergy
* Contraindication for ketamine infusion
* Contraindication for thoracic paravertebral block
* Anticipated postoperative positive pressure ventilation
* Body mass index more than 35
* Any known psychiatric disorder

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-09-25 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Postoperative morphine consumption | 24 hours postoperatively
  Amount of morphine (in milligrams) which is dispensed from a patient-controlled analgesia device (PCA)

SECONDARY OUTCOMES:
Time to first analgesia | 24 hours postoperatively
  Time period (in minutes) after the end of surgery until the time of first morphine solution is dispensed from PCA device
Peak flow rates (day 1) | 1 days
  The value of peak flow velocity obtained from the first postoperative day will be compare with the value at the preoperative period
Peak flow rates (day 2) | 2 days
  The value of peak flow velocity obtained from the first postoperative day will be compare with the value at the preoperative period
Chronic post-surgical pain | 1 month
  The score of the Thai version of PainDetect questionnaire will be obtained at 1 month postoperatively
Chronic post-surgical pain | 3 months
  The score of the Thai version of PainDetect questionnaire will be obtained at 3 months postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Sirilak Suksompong, Principal Investigator — Mahidol University
Locations (1):
- Siriraj Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gerner P. Postthoracotomy pain management problems. Anesthesiol Clin. 2008 Jun;26(2):355-67, vii. doi: 10.1016/j.anclin.2008.01.007. PMID 18456219
- [Background] Furrer M, Rechsteiner R, Eigenmann V, Signer C, Althaus U, Ris HB. Thoracotomy and thoracoscopy: postoperative pulmonary function, pain and chest wall complaints. Eur J Cardiothorac Surg. 1997 Jul;12(1):82-7. doi: 10.1016/s1010-7940(97)00105-x. PMID 9262085
- [Background] Agostini P, Cieslik H, Rathinam S, Bishay E, Kalkat MS, Rajesh PB, Steyn RS, Singh S, Naidu B. Postoperative pulmonary complications following thoracic surgery: are there any modifiable risk factors? Thorax. 2010 Sep;65(9):815-8. doi: 10.1136/thx.2009.123083. PMID 20805178
- [Background] Peng Z, Li H, Zhang C, Qian X, Feng Z, Zhu S. A retrospective study of chronic post-surgical pain following thoracic surgery: prevalence, risk factors, incidence of neuropathic component, and impact on qualify of life. PLoS One. 2014 Feb 28;9(2):e90014. doi: 10.1371/journal.pone.0090014. eCollection 2014. PMID 24587187
- [Background] Wildgaard K, Ringsted TK, Hansen HJ, Petersen RH, Werner MU, Kehlet H. Quantitative sensory testing of persistent pain after video-assisted thoracic surgery lobectomy. Br J Anaesth. 2012 Jan;108(1):126-33. doi: 10.1093/bja/aer325. Epub 2011 Oct 5. PMID 21980121
- [Background] Bertrand PC, Regnard JF, Spaggiari L, Levi JF, Magdeleinat P, Guibert L, Levasseur P. Immediate and long-term results after surgical treatment of primary spontaneous pneumothorax by VATS. Ann Thorac Surg. 1996 Jun;61(6):1641-5. doi: 10.1016/0003-4975(96)00190-7. PMID 8651762
- [Background] De Cosmo G, Aceto P, Gualtieri E, Congedo E. Analgesia in thoracic surgery: review. Minerva Anestesiol. 2009 Jun;75(6):393-400. Epub 2008 Oct 27. PMID 18953284
- [Background] Amlong C, Guy M, Schroeder KM, Donnelly MJ. Out-of-plane ultrasound-guided paravertebral blocks improve analgesic outcomes in patients undergoing video-assisted thoracoscopic surgery. Local Reg Anesth. 2015 Dec 15;8:123-8. doi: 10.2147/LRA.S86853. eCollection 2015. PMID 26730208
- [Background] Kaya FN, Turker G, Basagan-Mogol E, Goren S, Bayram S, Gebitekin C. Preoperative multiple-injection thoracic paravertebral blocks reduce postoperative pain and analgesic requirements after video-assisted thoracic surgery. J Cardiothorac Vasc Anesth. 2006 Oct;20(5):639-43. doi: 10.1053/j.jvca.2006.03.022. Epub 2006 Aug 8. PMID 17023279
- [Background] Suzuki M, Haraguti S, Sugimoto K, Kikutani T, Shimada Y, Sakamoto A. Low-dose intravenous ketamine potentiates epidural analgesia after thoracotomy. Anesthesiology. 2006 Jul;105(1):111-9. doi: 10.1097/00000542-200607000-00020. PMID 16810002